CLINICAL TRIAL: NCT02178800
Title: A Phase IIa Study to Evaluate the Safety, Tolerability and Pharmacokinetics of the Investigational Injectable HIV Integrase Inhibitor, GSK1265744, in HIV-uninfected Men and Women
Brief Title: Evaluating the Safety, Tolerability, and Pharmacokinetics of an Investigational, Injectable HIV Medicine (GSK1265744) in HIV-Uninfected Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HPTN 077; 11964 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Results first posted 2018-07-05 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: GSK1265744 (Experimental): Participants in Cohorts 1 and 2 will receive one GSK1265744 tablet orally every day from study entry through Week 4. They will then receive an injection of GSK1265744-at Weeks 5, 17, and 29 for participants in Cohort 1 and at Weeks 5, 9, 17, 25, and 33 for participants in Cohort 2.
  Interventions: Drug: GSK1265744 Tablets; Drug: Injectable GSK1265744
- Group 2: Placebo (Placebo Comparator): Participants in Cohorts 1 and 2 will receive one placebo tablet orally every day from study entry through Week 4. They will then receive an injection of placebo-at Weeks 5, 17, and 29 for participants in Cohort 1 and at Weeks 5, 9, 17, 25, and 33 for participants in Cohort 2.
  Interventions: Drug: Placebo for GSK1265744 Tablets; Drug: Injectable Placebo for GSK1265744

INTERVENTIONS:
Drug: GSK1265744 Tablets — 30-mg tablets, taken orally
  Other Names: Oral 744
  Arms: Group 1: GSK1265744
Drug: Injectable GSK1265744 — Cohort 1: 800-mg injection, administered as two 400-mg intramuscular (IM) gluteal injections
  Cohort 2: 600-mg injection, administered as one IM gluteal injection
  Other Names: GSK1265744 long acting; 744LA
  Arms: Group 1: GSK1265744
Drug: Placebo for GSK1265744 Tablets — Taken orally
  Arms: Group 2: Placebo
Drug: Injectable Placebo for GSK1265744 — Cohort 1: Sodium Chloride for Injection USP, 0.9%; administered as two 400-mg IM gluteal injections
  Cohort 2: Sodium Chloride for Injection USP, 0.9%; administered as one 600-mg IM gluteal injection
  Arms: Group 2: Placebo

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics (which is how the body interacts with drugs) of an investigational, injectable HIV medicine (GSK1265744) in healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
This study will evaluate GSK1265744, which is an investigational, injectable HIV medicine. The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of GSK1265744 in healthy, HIV-uninfected adults.

This study will enroll two cohorts of participants (Cohort 1 and Cohort 2). Within each cohort, participants will be randomly assigned to one of two groups: Group 1 will receive GSK1265744 tablets (also called oral 744) and injections (also called GSK1265744 long acting or 744LA), and Group 2 will receive placebo tablets and injections. Participants in Cohort 1 will attend several study visits through Week 81 or Week 105. Participants in Cohort 2 will attend several study visits through Week 85 or Week 109. From study entry through Week 4, participants in both cohorts will take a GSK1265744 tablet (Group 1) or a placebo tablet (Group 2) once a day. For 1 week after participants stop taking their assigned tablets, study researchers will assess safety and tolerability. If no safety or tolerability concerns are identified, participants will enter the injection phase of the study. Participants in Cohort 1 will receive two injections of GSK1265744 (Group 1) or placebo (Group 2) at Weeks 5, 17, and 29. Participants in Cohort 2 will receive one injection of GSK1265744 (Group 1) or placebo (Group 2) at Weeks 5, 9, 17, 25, and 33.

All study visits will include HIV counseling, a physical examination, a medical history review, and a blood collection. Select study visits will include adherence counseling, central nervous system (CNS) symptom assessment, behavioral and acceptability assessments, a urine collection, an electrocardiogram (ECG), and rectal and/or vaginal swabs.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 to 65 years old at the time of screening
* Willing to provide informed consent for the study
* In the last 12 months (at the time of screening):

  * No self-reported unprotected anal or vaginal intercourse with someone known to be HIV-infected or of unknown HIV infection status
  * No self-reported stimulant use (cocaine [including crack], methamphetamine, or non-physician-prescribed pharmaceutical-grade stimulants) or inhaled nitrate
  * No self-reported illicit injection drug use of any kind
  * No self-reported diagnosis of gonorrhea (GC), chlamydia (CT), incident syphilis, bacterial vaginosis, or trichomoniasis
  * Not reporting five or more different sexual partners, regardless of use of protection or knowledge of HIV status. More information on this criterion is available in the protocol.
* In general good health, as evidenced by the following laboratory values, which must be from specimens obtained within 45 days prior to study enrollment:

  * Non-reactive/negative HIV test results. More information on this criterion is available in the protocol.
  * Hemoglobin greater than 11 g/dL
  * Absolute neutrophil count greater than 750 cells/mm^3
  * Platelet count greater than or equal to 100,000/mm^3
  * Calculated creatinine clearance greater than or equal to 70 mL/minute using the Cockcroft-Gault equation
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to the upper limit of normal (ULN)
  * Total bilirubin less than or equal to Grade 1 and direct bilirubin less than or equal to ULN
  * Hepatitis B surface antigen (HBsAg) negative
  * Hepatitis C Ab negative
  * Note: Chemistry and hematology parameters which do not meet the inclusion criteria above may be repeated once during screening.
* No alcohol or substance use that, in the opinion of the study investigator, would interfere with the conduct of the study (e.g., provided by self-report, or found upon medical history and examination or in available medical records). More information on this criterion is available in the protocol.
* No medical condition that, in the opinion of the study investigator, would interfere with the conduct of the study (e.g., provided by self-report, or found upon medical history and examination or in available medical records)
* Willing to undergo all required study procedures

Additional requirements for all women:

* If of reproductive potential (defined as pre-menopausal women who have not had a sterilization procedure per self-report, such as hysterectomy, bilateral oophorectomy, tubal ligation, or salpingectomy), must have a negative urine pregnancy test performed (and results known) within 48 hours before initiating the protocol-specified medication(s) at enrollment. Women are considered menopausal if they have not had a menses for at least 12 months and have a follicle stimulating hormone (FSH) level of greater than 40 IU/L; if FSH testing is not available, they must have had amenorrhea for 24 or more consecutive months. (FSH testing is not a protocol requirement.)
* If of reproductive potential and participating in sexual activity that could lead to pregnancy, women must agree to use a form of contraception during the trial and for 30 days after stopping the oral study medication or for 52 weeks after stopping the long acting injectable from the list below:

  * Intrauterine device (IUD) or intrauterine system (IUS) that meets less than 1% failure rate as stated in the product label
  * Hormone-based contraceptive

Exclusion Criteria:

* One or more reactive or positive HIV test result at Screening or Enrollment, even if HIV infection is not confirmed
* Any active sexually transmitted infection detected by laboratory testing at Screening
* Co-enrollment in any other HIV interventional research study or other concurrent studies which may interfere with this study (as provided by self-report or other available documentation; exceptions may be made if appropriate after consultation with the Clinical Management Committee [CMC].)
* Past or current participation in HIV vaccine trial. An exception will be made for participants that can provide documentation of receipt of placebo (not active arm).
* Use of antiretroviral therapy (ART) (e.g., for non-occupational post-exposure prophylaxis [PEP] or PrEP) in the 90 days prior to study entry
* Clinically significant cardiovascular disease, including:
* ECG (one repeat ECG is allowed during screening; may be performed on the same day) with:

  * heart rate less than 45 or greater than 100 beats per minute for men, and less than 50 or greater than 100 beats per minute for women
  * interval from the beginning of the Q wave to the end of the S wave (QRS) duration greater than 120 msec
  * corrected QT (QTc) interval (B or F) greater than 450 msec
  * evidence of previous myocardial infarction (pathologic Q waves, S-T segment changes) (except early repolarization)
  * any clinically significant conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular [AV] block [2nd degree (type II) or higher], Wolf Parkinson White [WPW] syndrome) (any question of clinical significance should be referred to the CMC for adjudication)
  * sinus pauses greater than 3 seconds
  * any clinically significant arrhythmia that, in the opinion of the Investigator of Record (IoR) or designee, will interfere with the safety for the individual participant (any question of clinical significance should be referred to the CMC for adjudication)
  * or history of non-sustained (greater than or equal to 3 consecutive ventricular ectopic beats on ECG at screening or entry) or sustained ventricular tachycardia
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PTCA) or any clinically significant cardiac disease
* Systolic blood pressure at screening outside the range of 90 to 140 mm Hg or diastolic blood pressure outside the range of 45 to 90 mm Hg (confirmed on repeat measurement)
* Underlying skin disease or currently active skin disorder (e.g., infection, inflammation, dermatitis, eczema, psoriasis, urticaria). Mild cases of localized acne or folliculitis or other mild skin condition may not be exclusionary at the discretion of the IoR or designee in consultation with the CMC.
* Has a tattoo or other dermatological condition overlying the buttock region that in the opinion of the IoR or designee, in consultation with the CMC, may interfere with interpretation of injection site reactions
* Current or chronic history of liver disease (e.g., non-alcoholic or alcoholic steatohepatitis) or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome, asymptomatic gallstones, or cholecystectomy)
* Coagulopathy (primary or iatrogenic) that would contraindicate IM injection (concomitant anticoagulant or anti-platelet therapy use should be discussed with the CMC)
* Active or planned use of prohibited medications as described in the Investigator's Brochure or listed in the Study Specific Procedures (SSP) Manual (provided by self-report, or obtained from medical history or medical records)
* A score of greater than or equal to 8 on the WHO Alcohol Use Disorders Identification Test (AUDIT) at screening. Note: A score of greater than or equal to 8 indicates a medium to high level of problem alcohol use.
* For women: pregnant or currently breastfeeding, or intends to become pregnant and/or breastfeed during the study
* A history of seizure disorder, by self-report

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2015-02; Primary Completion 2017-04-05 (Actual); Study Completion 2018-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raphael J. Landovitz, MD, MSc, Study Chair — University of California, Los Angeles
Locations (8):
- United States (4):
  - UCLA CARE Center CRS, Los Angeles, California
  - Bridge HIV CRS, San Francisco, California
  - George Washington Univ. CRS, Washington D.C., District of Columbia
  - Chapel Hill CRS, Chapel Hill, North Carolina
- Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro, Brazil
- Malawi CRS, Lilongwe, Malawi
- South Africa (2):
  - Soweto HPTN CRS, Johannesburg, Gauteng
  - Vulindlela CRS, Durban, KwaZulu-Natal

REFERENCES:
- [Derived] Landovitz RJ, Li S, Eron JJ Jr, Grinsztejn B, Dawood H, Liu AY, Magnus M, Hosseinipour MC, Panchia R, Cottle L, Chau G, Richardson P, Marzinke MA, Eshleman SH, Kofron R, Adeyeye A, Burns D, Rinehart AR, Margolis D, Cohen MS, McCauley M, Hendrix CW. Tail-phase safety, tolerability, and pharmacokinetics of long-acting injectable cabotegravir in HIV-uninfected adults: a secondary analysis of the HPTN 077 trial. Lancet HIV. 2020 Jul;7(7):e472-e481. doi: 10.1016/S2352-3018(20)30106-5. Epub 2020 Jun 1. PMID 32497491
- [Derived] Landovitz RJ, Li S, Grinsztejn B, Dawood H, Liu AY, Magnus M, Hosseinipour MC, Panchia R, Cottle L, Chau G, Richardson P, Marzinke MA, Hendrix CW, Eshleman SH, Zhang Y, Tolley E, Sugarman J, Kofron R, Adeyeye A, Burns D, Rinehart AR, Margolis D, Spreen WR, Cohen MS, McCauley M, Eron JJ. Safety, tolerability, and pharmacokinetics of long-acting injectable cabotegravir in low-risk HIV-uninfected individuals: HPTN 077, a phase 2a randomized controlled trial. PLoS Med. 2018 Nov 8;15(11):e1002690. doi: 10.1371/journal.pmed.1002690. eCollection 2018 Nov. PMID 30408115

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: GSK1265744: Participants in Cohorts 1 and 2 will receive one GSK1265744 tablet orally every day from study entry through Week 4. They will then receive an injection of GSK1265744-at Weeks 5, 17, and 29 for participants in Cohort 1 and at Weeks 5, 9, 17, 25, and 33 for participants in Cohort 2.
  GSK1265744 Tablets: 30-mg tablets, taken orally
  Injectable GSK1265744: Cohort 1: 800-mg injection, administered as two 400-mg intramuscular (IM) gluteal injections
  Cohort 2: 600-mg injection, administered as one IM gluteal injection
- Group 2: Placebo: Participants in Cohorts 1 and 2 will receive one placebo tablet orally every day from study entry through Week 4. They will then receive an injection of placebo-at Weeks 5, 17, and 29 for participants in Cohort 1 and at Weeks 5, 9, 17, 25, and 33 for participants in Cohort 2.
  Placebo for GSK1265744 Tablets: Taken orally
  Injectable Placebo for GSK1265744: Cohort 1: Sodium Chloride for Injection USP, 0.9%; administered as two 400-mg IM gluteal injections
  Cohort 2: Sodium Chloride for Injection USP, 0.9%; administered as one 600-mg IM gluteal injection
Period: Overall Study
Arm/Group | Group 1: GSK1265744 | Group 2: Placebo
Started | 151 | 48
Completed | 131 (Number of participants who weren't terminated at week 41) | 42 (Number of participants who weren't terminated at week 41)
Not Completed | 20 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: GSK1265744 | Group 2: Placebo | Total
Number analyzed (Participants) | 151 | 48 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (11.4) | 35 (11.0) | 33 (11.3)
Age, Customized [Count of Participants; unit: Participants]
  18 - 25 | 52 | 9 | 61
  26 - 35 | 53 | 17 | 70
  36 - 45 | 21 | 14 | 35
  46 - 55 | 15 | 4 | 19
  56 - 65 | 10 | 4 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 32 | 132
  Male | 51 | 16 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Latino | 36 | 11 | 47
  Non-hispanic Asian | 3 | 2 | 5
  Non-hispanic Black | 64 | 18 | 82
  Non-hispanic White | 42 | 12 | 54
  Non-hispanic mixed/other | 6 | 5 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 80 | 26 | 106
  Malawi | 14 | 3 | 17
  Brazil | 24 | 10 | 34
  South Africa | 33 | 9 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Any Grade 2 or Higher Clinical Adverse Events (AEs) and Laboratory Abnormalities That Occur From the Initial Injection to Week 41 Among Participants Who Receive at Least One Injection (Injectable Phase Only)
Description: An adverse events (AE) or laboratory abnormality can be an unfavorable or unintended sign, symptom or disease temporally associated with the use of an investigational product, whether or not considered related to the product. AE severity was graded per the DAIDS Table for Grading Adult and Pediatric Adverse Events, Version 2.0, November 2014. The outcome in this table is stratified by arm.
Time Frame: Measured through Week 41
Population: This population includes participants who receive at least one injection in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: GSK1265744 | Group 2: Placebo
Number analyzed (Participants) | 134 | 43
Participants | 121 | 38

2. Primary Outcome: Number of Participants Who Discontinue Injectable Study Product for Reasons of Toxicity, Tolerability, or Acceptability That Occur From the Initial Injection to Week 41 Among Participants Who Receive at Least One Injection (Injectable Phase Only)
Description: Stratified by arm
Time Frame: Measured through Week 41
Population: This population includes participants who received at least one injection in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: GSK1265744 | Group 2: Placebo
Number analyzed (Participants) | 134 | 43
Participants | 11 | 2

3. Primary Outcome: Plasma Drug Levels of GSK1265744 at Designated Time Points After Each Injection of 744LA (Injectable Formulation of GSK1265744)
Description: Geometric means and 90% prediction intervals by sex at birth and cohort are reported.
Time Frame: Measured through Week 41
Population: PK sample size varies by visit due to reasons such as missing visits, different schedule and sample contamination.
Measure: Geometric Mean (90% Confidence Interval); unit: ug/ml
Groups:
- Female, Cohort 1: Female, GSK1265744 arm, Cohort 1 participants who received at least one injection only. Plasma drug concentrations at Week 6, 9,13,17,18,23,29,30,35 and 41 are measured.
- Male, Cohort 1: Male, GSK1265744 arm, Cohort 1 participants who received at least one injection only. Plasma drug concentrations at Week 6, 9,13,17,18,23,29,30,35 and 41 are measured.
- Female, Cohort 2: Female, GSK1265744 arm, Cohort 2 participants who received at least one injection only. Plasma drug concentrations at Week 6, 9,10,13,17,18,21,25,26,29,33,34,37 and 41 are measured.
- Male, Cohort 2: Male, GSK1265744 arm, Cohort 2 participants who received at least one injection only. Plasma drug concentrations at Week 6, 9,10,13,17,18,21,25,26,29,33,34,37 and 41 are measured.
Arm/Group | Female, Cohort 1 | Male, Cohort 1 | Female, Cohort 2 | Male, Cohort 2
Number analyzed (Participants) | 49 | 25 | 40 | 20
ug/ml
  Week 6 | 1.32 [0.49 to 3.54] | 2.40 [0.63 to 9.22] | 1.29 [0.33 to 5.05] | 2.28 [0.67 to 7.72]
  Week 9: number analyzed (Participants) | 49 | 25 | 39 | 20
  Week 9 | 1.49 [0.53 to 4.18] | 1.77 [0.70 to 4.47] | 1.31 [0.38 to 4.44] | 1.79 [0.93 to 3.44]
  Week 10: number analyzed (Participants) | 0 | 0 | 39 | 20
  Week 10 |  |  | 2.56 [0.94 to 6.98] | 3.58 [1.42 to 9.00]
  Week 13: number analyzed (Participants) | 49 | 25 | 39 | 20
  Week 13 | 1.18 [0.52 to 2.69] | 0.90 [0.40 to 2.01] | 2.24 [0.89 to 5.65] | 2.55 [1.22 to 5.33]
  Week 17: number analyzed (Participants) | 49 | 25 | 39 | 20
  Week 17 | 0.95 [0.42 to 2.14] | 0.49 [0.19 to 1.31] | 1.82 [0.79 to 4.21] | 1.29 [0.54 to 3.09]
  Week 18: number analyzed (Participants) | 40 | 23 | 38 | 20
  Week 18 | 2.11 [0.94 to 4.75] | 2.33 [0.72 to 7.53] | 3.09 [1.32 to 7.25] | 2.73 [1.03 to 7.29]
  Week 21: number analyzed (Participants) | 0 | 0 | 38 | 20
  Week 21 |  |  | 2.74 [1.29 to 5.79] | 2.07 [0.87 to 4.90]
  Week 23: number analyzed (Participants) | 40 | 23 | 0 | 0
  Week 23 | 2.02 [0.86 to 4.74] | 1.48 [0.84 to 2.59] |  |
  Week 25: number analyzed (Participants) | 0 | 0 | 37 | 20
  Week 25 |  |  | 2.00 [0.96 to 4.16] | 1.11 [0.38 to 3.20]
  Week 26: number analyzed (Participants) | 0 | 0 | 38 | 20
  Week 26 |  |  | 3.07 [1.30 to 7.27] | 2.84 [1.24 to 6.49]
  Week 29: number analyzed (Participants) | 39 | 23 | 38 | 20
  Week 29 | 1.37 [0.61 to 3.06] | 0.78 [0.30 to 2.02] | 2.68 [1.23 to 5.81] | 2.17 [0.98 to 4.81]
  Week 30: number analyzed (Participants) | 35 | 23 | 0 | 0
  Week 30 | 2.78 [1.23 to 6.28] | 3.48 [1.43 to 8.48] |  |
  Week 33: number analyzed (Participants) | 0 | 0 | 36 | 19
  Week 33 |  |  | 2.10 [0.94 to 4.70] | 1.50 [0.55 to 4.11]
  Week 34: number analyzed (Participants) | 0 | 0 | 35 | 19
  Week 34 |  |  | 3.59 [1.50 to 8.58] | 3.60 [1.48 to 8.74]
  Week 35: number analyzed (Participants) | 35 | 23 | 0 | 0
  Week 35 | 2.41 [1.03 to 5.61] | 1.85 [1.07 to 3.20] |  |
  Week 37: number analyzed (Participants) | 0 | 0 | 36 | 18
  Week 37 |  |  | 2.73 [1.06 to 7.06] | 2.71 [1.67 to 4.40]
  Week 41: number analyzed (Participants) | 36 | 22 | 35 | 18
  Week 41 | 1.68 [0.78 to 3.62] | 0.82 [0.27 to 2.54] | 2.06 [0.77 to 5.49] | 1.68 [0.68 to 4.17]

4. Secondary Outcome: Number of Participants Experiencing Grade 2 or Higher Clinical Adverse Events (AEs) and Laboratory Abnormalities During Tail Phase
Description: as for outcome 1
Time Frame: Measured from 12 weeks after last injection through Week 105 for Cohort 1 and 8 weeks after last injection through Week 109 for Cohort 2
Population: This includes participants who entered tail phase
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: GSK1265744 | Group 2: Placebo
Number analyzed (Participants) | 130 | 42
Participants | 107 | 18

5. Secondary Outcome: Number of Participants Experiencing Grade 2 or Higher Clinical Adverse Events (AEs) and Laboratory Abnormalities Prior to Completion of the Oral Phase
Description: as for outcome 1
Time Frame: Measured through Week 5
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: GSK1265744 | Group 2: Placebo
Number analyzed (Participants) | 151 | 48
Participants | 84 | 25

6. Secondary Outcome: Number of Participants Willing to Use an Injectable Agent Such as the Study Product for HIV Prevention in the Future
Description: Stratified by Visit and Cohort
Time Frame: Measured from week 6 through Week 30 in cohort 1 and Week 34 in cohort 2
Population: Sample size varies by visit due to reasons such as missing visits and different schedules.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Participants who were planned to receive IM injections of 744LA or placebo at three time points at 12 week intervals.Two sequential 400 mg gluteal injections were given at each injection visit (if not discontinued).
- Cohort 2: participants who were planned to receive IM injections of 744LA or placebo at five time points at 4 and 8 week intervals.One 600 mg gluteal injection was given at each injection visit (if not discontinued).
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 98 | 78
Participants
  Week 6 | 80 | 74
  Week 10: number analyzed (Participants) | 0 | 77
  Week 10 |  | 74
  Week 18: number analyzed (Participants) | 88 | 75
  Week 18 | 81 | 73
  Week 26: number analyzed (Participants) | 0 | 75
  Week 26 |  | 71
  Week 30: number analyzed (Participants) | 77 | 0
  Week 30 | 69 |
  Week 34: number analyzed (Participants) | 0 | 70
  Week 34 |  | 65

7. Secondary Outcome: Number of Participants With HIV Infections Through the Study Period, Stratified by Arm
Time Frame: Measured through Week 105 for Cohort 1 and Week 109 for Cohort 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: GSK1265744 | Group 2: Placebo
Number analyzed (Participants) | 151 | 48
Participants | 1 | 0

8. Secondary Outcome: Self-reported Sexual Behavior (Number of Sexual Partners) During the Study Period
Description: Week 29/31 is a combination of week 29, cohort 1 and week 33, cohort 2. The outcome in this table is stratified by arm.
Time Frame: Measured through Week 77
Population: Analysis sample size is different at each visit due to multiple reasons (early termination, missing data, study unblinding, etc.)
Measure: Mean (Standard Deviation); unit: partners
Arm/Group | Group 1: GSK1265744 | Group 2: Placebo
Number analyzed (Participants) | 151 | 48
partners
  Enrollment Visit | 0.81 (0.46) | 0.92 (0.65)
  Week 5: number analyzed (Participants) | 134 | 45
  Week 5 | 0.84 (0.44) | 0.78 (0.67)
  Week 17: number analyzed (Participants) | 132 | 43
  Week 17 | 0.81 (0.54) | 0.84 (0.57)
  Week 29/33: number analyzed (Participants) | 125 | 41
  Week 29/33 | 0.85 (0.57) | 0.80 (0.46)
  Week 41: number analyzed (Participants) | 130 | 42
  Week 41 | 0.85 (0.66) | 0.88 (0.45)
  Week 53: number analyzed (Participants) | 129 | 41
  Week 53 | 0.84 (0.62) | 0.83 (0.50)
  Week 65: number analyzed (Participants) | 115 | 33
  Week 65 | 0.87 (0.76) | 0.88 (0.48)
  Week 77: number analyzed (Participants) | 110 | 22
  Week 77 | 0.84 (0.61) | 0.82 (0.50)

9. Secondary Outcome: Number of Injectable Hormonal-contraception-using Female Participants Experiencing Grade 2 or Higher Clinical AE and Laboratory Abnormalities During Oral Phase
Description: as for outcome 1
Time Frame: Measured through Week 4
Population: This population includes injectable hormonal-contraception-using female participants in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: GSK1265744 | Group 2: Placebo
Number analyzed (Participants) | 34 | 13
Participants | 17 | 7

10. Secondary Outcome: Number of Injectable Hormonal-contraception-using Female Participants Experiencing Grade 2 or Higher Clinical AE and Laboratory Abnormalities During Injection Phase
Time Frame: Measured from first injection through 12 weeks after last injection for Cohort 1 and 8 weeks after last injection for Cohort 2
Population: This population includes injectable hormonal-contraception-using female participants who received at least one injection of study drug in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: GSK1265744 | Group 2: Placebo
Number analyzed (Participants) | 32 | 12
Participants | 29 | 12

11. Secondary Outcome: Number of Injectable Hormonal-contraception-using Female Participants Who Discontinue Study Product for Reasons of Toxicity, Tolerability, or Acceptability During Oral Phase
Description: Stratified by arm
Time Frame: Measured through Week 4
Population: This population includes injectable hormonal-contraception-using female participants in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: GSK1265744 | Group 2: Placebo
Number analyzed (Participants) | 34 | 13
Participants | 0 | 0

12. Secondary Outcome: Number of Injectable Hormonal-contraception-using Female Participants Who Discontinue Study Product for Reasons of Toxicity, Tolerability, or Acceptability During Injection Phase
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: GSK1265744 | Group 2: Placebo
Number analyzed (Participants) | 32 | 12
Participants | 3 | 0

13. Secondary Outcome: Number of Participants Who Discontinue Oral Study Product for Reasons of Toxicity, Tolerability, or Acceptability Prior to Completion of the Oral Phase
Description: Stratified by arm
Time Frame: Measured through Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: GSK1265744 | Group 2: Placebo
Number analyzed (Participants) | 151 | 48
Participants | 6 | 0

ADVERSE EVENTS:
Time Frame: 41 weeks
Arm/Group | Group 1: GSK1265744 | Group 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/48
Serious Adverse Events (participants affected / at risk) | 4/151 | 2/48
Other Adverse Events (participants affected / at risk) | 147/151 | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: GSK1265744 (N=151) | Group 2: Placebo (N=48)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Sensory loss (Nervous system disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Laryngitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: GSK1265744 (N=151) | Group 2: Placebo (N=48)
Abdominal discomfort (Gastrointestinal disorders) | 2 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (9) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 8 (12) | 4 (4)
Abnormal loss of weight (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 18 (26) | 5 (8)
Allergic pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Amylase decreased (Investigations) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 18 (32) | 5 (10)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (2) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (13) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 13 (18) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (18) | 3 (3)
Bacterial vaginosis (Infections and infestations) | 3 (3) | 2 (2)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Bilirubin conjugated increased (Investigations) | 7 (10) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Blood bicarbonate decreased (Investigations) | 24 (43) | 10 (18)
Blood bilirubin increased (Investigations) | 3 (5) | 3 (5)
Blood calcium decreased (Investigations) | 9 (10) | 4 (8)
Blood calcium increased (Investigations) | 5 (5) | 3 (3)
Blood cholesterol increased (Investigations) | 5 (5) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 25 (37) | 8 (14)
Blood creatinine increased (Investigations) | 19 (33) | 4 (6)
Blood glucose decreased (Investigations) | 29 (56) | 11 (19)
Blood glucose increased (Investigations) | 56 (99) | 21 (39)
Blood magnesium decreased (Investigations) | 18 (31) | 8 (11)
Blood magnesium increased (Investigations) | 2 (2) | 0 (0)
Blood phosphorus decreased (Investigations) | 25 (38) | 10 (17)
Blood potassium decreased (Investigations) | 8 (11) | 1 (1)
Blood potassium increased (Investigations) | 3 (3) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 7 (9) | 1 (1)
Blood pressure systolic increased (Investigations) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 8 (9) | 1 (1)
Blood sodium increased (Investigations) | 8 (11) | 3 (3)
Blood triglycerides increased (Investigations) | 7 (7) | 1 (1)
Body tinea (Infections and infestations) | 6 (6) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (2) | 0 (0)
Breast cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Carbon dioxide decreased (Investigations) | 8 (15) | 3 (5)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Cervicitis (Infections and infestations) | 0 (0) | 1 (1)
Chemical burn of skin (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest pain (General disorders) | 5 (5) | 0 (0)
Chikungunya virus infection (Infections and infestations) | 2 (2) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Chlamydial infection (Infections and infestations) | 2 (2) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Complication of device insertion (General disorders) | 1 (1) | 0 (0)
Complication of device removal (General disorders) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 7 (8) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 2 (2) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 2 (2) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (6) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 6 (7) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 71 (168) | 21 (47)
Cutaneous sporotrichosis (Infections and infestations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Device breakage (Product Issues) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 13 (16) | 6 (10)
Disturbance in attention (Nervous system disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 22 (28) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 4 (4) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 3 (4)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Electrocardiogram PR prolongation (Investigations) | 3 (4) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 7 (13) | 3 (4)
Electrocardiogram T wave inversion (Investigations) | 1 (1) | 1 (2)
Electrocardiogram repolarisation abnormality (Investigations) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Essential hypertension (Vascular disorders) | 1 (3) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 11 (15) | 6 (7)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 1 (1)
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 4 (4) | 0 (0)
Fungal infection (Infections and infestations) | 2 (2) | 0 (0)
Fungal skin infection (Infections and infestations) | 2 (2) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 5 (5) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (5) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 6 (6) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0)
Genital candidiasis (Infections and infestations) | 2 (3) | 0 (0)
Genital herpes (Infections and infestations) | 1 (1) | 0 (0)
Genital infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Genitourinary tract gonococcal infection (Infections and infestations) | 2 (2) | 0 (0)
Gingivitis (Infections and infestations) | 3 (3) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 6 (11) | 1 (3)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 53 (78) | 11 (13)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Human bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hunger (General disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperphagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 3 (3) | 1 (1)
Hypersomnia (Nervous system disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 8 (8) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 7 (10) | 1 (1)
Hypobarism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (12) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (8) | 1 (2)
Implant site pain (General disorders) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Induration (General disorders) | 2 (2) | 0 (0)
Infected bite (Infections and infestations) | 2 (2) | 0 (0)
Infection parasitic (Infections and infestations) | 2 (2) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 10 (11) | 4 (5)
Influenza like illness (General disorders) | 15 (19) | 1 (1)
Initial insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Injection related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 19 (23) | 2 (2)
Injection site dermatitis (General disorders) | 1 (1) | 0 (0)
Injection site discomfort (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 10 (16) | 0 (0)
Injection site induration (General disorders) | 24 (39) | 1 (2)
Injection site nodule (General disorders) | 7 (9) | 0 (0)
Injection site pain (General disorders) | 120 (567) | 11 (29)
Injection site pruritus (General disorders) | 4 (6) | 0 (0)
Injection site reaction (General disorders) | 4 (5) | 0 (0)
Injection site swelling (General disorders) | 11 (17) | 0 (0)
Injection site warmth (General disorders) | 3 (4) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 13 (18) | 2 (2)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Laryngitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Ligament laxity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Lipase increased (Investigations) | 23 (34) | 14 (26)
Low density lipoprotein increased (Investigations) | 9 (9) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 2 (3) | 0 (0)
Metabolic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Molluscum contagiosum (Infections and infestations) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 (14) | 4 (5)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 16 (19) | 4 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 8 (8) | 4 (7)
Nausea (Gastrointestinal disorders) | 18 (23) | 5 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (3) | 1 (2)
Night blindness (Eye disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 0 (0)
Oligomenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 2 (2) | 1 (1)
Oropharyngeal gonococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis media bacterial (Infections and infestations) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10) | 2 (2)
Papule (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 7 (9) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 2 (2)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 2 (2) | 0 (0)
Penile ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal exudate (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis bacterial (Infections and infestations) | 3 (4) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (3) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (2) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Proctitis chlamydial (Infections and infestations) | 1 (1) | 0 (0)
Protein urine (Investigations) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 5 (5) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Pseudopapilloedema (Eye disorders) | 1 (1) | 0 (0)
Puncture site pain (General disorders) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 9 (10) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rhinitis (Infections and infestations) | 3 (3) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Schistosomiasis (Infections and infestations) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1)
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 3 (3) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 5 (6) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 2 (2) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Somnolence (Nervous system disorders) | 3 (3) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 2 (2) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 1 (1)
Testicular swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 1 (2) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 1 (1)
Tinea versicolour (Infections and infestations) | 2 (2) | 0 (0)
Tongue coated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 3 (3) | 1 (1)
Tonsillitis bacterial (Infections and infestations) | 4 (4) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 3 (3) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Trichoglossia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 25 (41) | 11 (13)
Upper respiratory tract infection bacterial (Infections and infestations) | 10 (13) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urethritis gonococcal (Infections and infestations) | 1 (1) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 9 (11) | 2 (2)
Urinary tract infection bacterial (Infections and infestations) | 7 (9) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (8) | 2 (2)
Urticaria papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 5 (5) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 5 (5) | 2 (3)
Viral pharyngitis (Infections and infestations) | 5 (5) | 0 (0)
Viral rhinitis (Infections and infestations) | 6 (9) | 0 (0)
Viral tonsillitis (Infections and infestations) | 1 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 16 (18) | 8 (10)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 9 (14) | 2 (3)
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 6 (6) | 1 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 3 (4) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vulvovaginitis (Infections and infestations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 2 (4) | 3 (4)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0)
Xerosis (General disorders) | 1 (1) | 0 (0)
Zika virus infection (Infections and infestations) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-10-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT02178800/Prot_001.pdf
  • Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT02178800/SAP_000.pdf